CLINICAL TRIAL: NCT04640324
Title: The Role of the PNPLA3, TM6SF2 and MBOAT7 Genetic Variants in the Response to Silybin-phospholipid Complex, Vitamin D and Vitamin E Based Therapy for Non-alcoholic Fatty Liver Disease Patients
Brief Title: Effect of PNPLA3, TM6SF2 and MBOAT7 Genetic Variants on Non-alcoholic Fatty Liver Disease Therapeutic Outcome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Federico II University (Other); University of Salerno (Other)
Responsible Party: Principal Investigator, Alessandro Federico, Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 531/2016
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Insulin Resistance
Keywords: non-alcoholic fat ty liver disease; genetics; insulin resistance; nutraceutics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The 92 enrolled patients were divided in three groups: NAFLD wild type control group (n. 30), NAFLD treated wild type group (n. 30), NAFLD treated mutated group (n. 32). The block randomization method was used to randomize the 60 not mutated patients in the NAFLD wild-type control group and NAFLD treated wild type one.
  The patients inserted in the NAFLD treated wild type and NAFLD treated mutated groups were undergone to an oral administration of 303mg of silybin-phospholipid complex, 10mg of vitamin D, and 15mg of vitamin E, twice a day for six months. At the baseline and end of treatment, the assessment of WHtR, blood pressure measurement, BMI, Blood glucose and insulin, HOMA-IR, AST, ALT, GGT, blood count, CRP, TBARS, liver stiffness and CAP was performed. During the experimental observation, patients were on free diet on the basis of dietary habits before the enrollment and any type of physical exercise was recommended during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NAFLD wild type control group (No Intervention): Consisted of not treated NAFLD wild type patients
- NAFLD wild type treated group (Active Comparator): Consisted of NAFLD wild type patients treated with oral administration of 303mg of silybin-phospholipid complex, 10mg of vitamin D, and 15mg of vitamin E, twice a day six months
  Interventions: Drug: Nutraceutical therapy
- NAFLD mutated treated group (Experimental): Consisted of NAFLD patients carrying at least one mutation among PNPLA3, TM6SF2, MBOAT7 genes, treated with oral administration of 303mg of silybin-phospholipid complex, 10mg of vitamin D, and 15mg of vitamin E, twice a day six months
  Interventions: Drug: Nutraceutical therapy

INTERVENTIONS:
Drug: Nutraceutical therapy — Oral administration of 303mg of silybin-phospholipid complex, 10mg of vitamin D, and 15mg of vitamin E, twice a day for six months
  Other Names: Silybin-phospholipid, Vitamin D and vitamin E complex
  Arms: NAFLD mutated treated group; NAFLD wild type treated group

SUMMARY:
Patatin-like phospholipase domain-containing protein-3 (PNPLA3), the transmembrane 6 superfamily member 2 protein (TM6SF2) and membrane bound O-acyltransferase domain containing 7 (MBOAT7) genes are involved in non-alcoholic fatty liver disease (NAFLD) development and worsening. Following the actual scientific knowledge, some studies have identified the genetic background surrounding NAFLD, counting up to forty different genetic variants that seem to exert also a crucial role in the disease evolution, according to the natural history, until hepatocellular carcinoma onset. However, few data exist regarding their influence on the treatment response. The aim was to explore the effect of 303 mg of silybin-phospholipids complex, 10 mg of vitamin-D and 15 mg of vitamin-E twice a day for six months in NAFLD patients carrying PNPLA3-rs738409, TM6SF2-rs58542926 and MBOAT7-rs641738 genetic variants. The assessed mutations are independently associated with no response to a silybin/vitamin D-based therapy and could be useful therapeutic predictive markers in this context.

DETAILED DESCRIPTION:
The aim of this study was to evaluate if the PNPLA3 rs738409, TM6SF2 rs58542926 and MBOAT7 rs641738 could influence the response of NAFLD patients regarding metabolic parameters, liver damage and hepatic fat accumulation ones, to a treatment with 303 mg of silybin-phospholipids complex, 10 mg of vitamin D, and 15 mg of vitamin E twice a day for six months.

The investigators performed a baseline comparison of Weight, waist-to-height ratio (WHtR), blood pressure measurement, body mass index (BMI), Blood glucose and insulin, the homeostatic model for insulin resistance assessment (HOMA-IR), aspartate and alanine aminotransferase (AST, ALT), gamma-glutamyl transferase (GGT), blood count, C reactive protein (CRP), the Thiobarbituric Acid Reactive Substance (TBARS), liver stiffness and controlled attenuation parameter (CAP) among the three study groups: NAFLD wild type control group (n. 30), NAFLD treated wild type group (n. 30), NAFLD treated mutated group (n. 32). The block randomization method was used to randomize the 60 not mutated patients in the NAFLD wild-type control group and NAFLD treated wild type one, using the online randomization software http://www.graphpad.com/quickcalcs/index.cfm.

The wild-type control group was composed by NAFLD patients without PNPLA3, TM6SF2 and MBOAT7 mutations that did not receive any type of treatment during the study period.

The patients inserted in the NAFLD treated wild type and NAFLD treated mutated groups were undergone to an oral administration of 303mg of silybin-phospholipid complex, 10mg of vitamin D, and 15mg of vitamin E, twice a day for six months. None of the enrolled patients dropped-out the study.

At the end of treatment, the assessment of WHtR, blood pressure measurement, BMI, Blood glucose and insulin, HOMA-IR, AST, ALT, GGT, blood count, CRP, TBARS, liver stiffness and CAP was re-performed. During the experimental observation, patients were on free diet on the basis of dietary habits before the enrollment and any type of physical exercise was recommended during the study period. Food intake was evaluated both at baseline and end of treatment using a computerized software. The investigators recorded, with a diet diary, the food intake of a complete week, including working days and the weekend. On the basis of the quantities and qualities of food consumed, the soft elaborates the daily energy intake and the percentage/caloric amount of macronutrients. For the physical exercise assessment, the investigators submitted a specific questionnaire at baseline and end of treatment with some simple questions: Are the participant doing or have the participant ever done (in the last two years) sport in a continuative and regular way? Have the participant changed his/her daily physical activity in the last six months? 1: no, 2: yes; if yes, has the physical activity enhanced or worsened? Alcohol consumption was assessed at the beginning and at the end of the treatment. One hundred two patients with histological diagnosis of NAFLD followed by the Hepatogastroenterology Division of the University of Campania "Luigi Vanvitelli, between January and October 2017 were screened, after signing an informed consent, for the PNPLA3 rs738409, TM6SF2 rs58542926 and MBOAT7 rs641738 genetic variants and thirty-two met the inclusion criteria for the study and showed at least one among PNPLA3 I148I/M, I148M/M, TM6SF2 167E/K, 167K/K and MBOAT7 TMC4C/T or TMC4T/T genetic variants, were enrolled together with sixty patients without the mutations. Ten patients were excluded from the enrollment due to the coexistence of several comorbidities and/or advanced stages liver disease such as cirrhosis and/or hepatocellular carcinoma (HCC).

The definition of the presence/absence of NAFLD and the staging were assessed by performing a liver biopsy, serological tests and collecting clinical data. Medical history, alcohol consumption (AUDIT-C), medications, drug abuse, smoking habits, were also investigated. Blood pressure, weight, height were directly measured and WHtR was calculated. BMI was also calculated by dividing the weight (kg) by the square of height (m). The patients were undergone after 12 hours fast to peripheral venous blood samples collection in order to evaluate some biochemical parameters and to perform the genetic analysis.

Insulin, GGT, CRP, levels were measured enzymatically using commercially available kits, AST, ALT and glucose using colorimetric assay kit (Amplite 13801/13803 and Thermo Fisher Scientific EIAGLUC). HOMA-IR was also calculated using the formula: fasting insulin (μU/mL) × plasma glucose (mmol/L)/22.5.

FibroScan® transient elastography (TE) was performed using the FibroScan® version 502 (Echosens, Paris, France) with standard probes (M and XL probes. The extra large (XL) probe was used when the distance from the skin to the liver capsule, assessed by ultrasonography, exceeded 2.5 cm and/or when BMI was >30. FibroScan® was performed by an expert physician obtaining ten acceptable measurements, defined as a successful liver stiffness (LS) measurement, with the maximum number of attempts set at 20. The criteria proposed by Boursier et al. were used to consider the measurement "very reliable" (IQR/M ≤ 0:1), "reliable" (0:1 < IQR/M ≤ 0:3 or IQR/M > 0:3 with LS median < 7:1 kPa), or "poorly reliable" (IQR/M > 0:3 with LS median ≥ 7:1 kPa). On the basis of CAP these scores, the investigators classified the enrolled patients in S0, no steatosis (0%-10% fat; 0-237 dB/m); S1, mild steatosis (11%-33% fat; 238-259 dB/m); S2, moderate steatosis (34%-66% fat; 260-292 dB/m); and S3, severe steatosis (>67% fat; ≥293 dB/m) in accordance with calculation of the attenuation of ultrasonic signals used for TE.

TBARS assay was performed using 10 μl of serum. The cromogen TBARS was quantified using a spectrophotometer at a wavelength of 532nm with 1,1,3,3-tetramethoxyprophane as a standard. The amount of TBARS was expressed as nmol/μg of protein. Presented data are the mean ± standard deviation, resulting from three independent experiments.

The genomic DNA extraction from peripheral blood samples was performed by using the extraction kit PureLink Genomic DNA Kit (Invitrogen by Life Technologies, USA). The DNA amount of each sample was assessed by spectrophotometer (NanoDrop Thermo Fisher Scientific) using a wave length of 260 nm. The presence of sample contamination was assessed by using a 280 nm wave length evaluation and all the sample showed good degree of purity because of the 260/280 ratio was between 1.8 and 2. The DNA extracted was then stored in -20°C freezer until the analysis of the polymorphisms.

The single nucleotide polymorphisms (SNPs) analysis, using the access code to the data bank TM6SF2 rs58542926 (SNP 1), MBOAT7 rs641738 (SNP2), PNPLA3 rs738409 (SNP3), was performed using the DNA genotyping RealTime PCR with TaqMan (Applied Biosystem) c_89463510_10 for SNP 1, c_8716820_10 for SNP 2, c_7241_10 for SNP 3 probes. All the evaluations were done in three phases: DNA PCR amplification, allelic identification and end point analysis with melting curve.

The first phase was done by using the AmpliTaq Gold® DNA polymerase contained in the TaqMan Universal PCR Master Mix amplifying the target sequence by specific primers contained in the SNP Genotyping Assay 40X together with TaqMan® MGB probes: one marked with fluorochrome VIC® that recognize the sequence of the allele 1 and another probe marked with fluorochrome FAM™ that recognize the sequence of the allele 2. For each experiment a 48 well plate was used, in which, a part of the biologic samples of unknown genotype for the SNP analysis, three different negative controls were analyzed in order to avoid possible errors due to the contamination of samples. Each experiment was done in triplicate. The amplifications were performed using the StepOne™ Real Time PCR System (Applied Biosystems). The genotyping assessment is based on the allelic discrimination thanks to a different fluorescence of the specific gene primer, using two MGB TaqMan® probes, marked at 5' with a different fluorochrome: SNP1 in reverse G in VIC® and A in FAM™; SNIP2 in forward C in VIC® and T in FAM™; SNIP3 in forward C in VIC® e G in FAM™. For the results analysis the software StepOne™2.0 was used. After the differentiation of the fluorescence made from the probes to the background in each well, it measures the normalized signal intensities (Rn) projecting the results in allelic discrimination plot. The software gives to the samples a specific genotype based on the fluorescence signal position: horizontal axis (allele one), vertical axis (allele 2) diagonal axis (both allele one and two). The prevalence of a specific fluorescence on the other one identified the homozygosis genotype, on the contrary the presence of both the heterozygosis.

Statistical Analysis The number of patients (30 in the NAFLD wild-type control group, 30 in the NAFLD treated wild type and 32 in NAFLD treated mutated ones) was calculated using the power and sample size calculation function of STATA-14® for mac-OS, on the basis of an expected difference among the study groups in the response of the HOMA-IR to the therapy, assuming a double amount of patient responder to the therapy in wild type group in comparison to the mutated one. Specifically, the investigators considered the patients responder if at least one of the following criteria was addressed: normalization of the HOMA-IR (<2.5) at the end of treatment starting from baseline values greater than 2.5; reduction of the HOMA-IR ≥ 2 points at the end of treatment in comparison to baseline. On the basis of this difference, the investigators estimated 29 patients per arm as the correct sample size of subjects to be investigate maintaining an 0.01 alpha error and a 90% statistical power in a two-sided test with a 95% Confidence Interval. A Kolgoromov-Smirnov for normality was performed to evaluate if parametric or non-parametric analysis should be applied. Wilcoxon signed ranks test, Mann-Whitney U test and t-test for dependent or independent groups were performed in order to compare continuous variables. The Kruskal-Wallis test or ANOVA test with post-hoc Bonferroni analysis, in case of non-normal or normal distribution respectively, were performed to compare the continuous variables among three groups. Pearson's or Kendall Tau-b correlations as well as linear regression were applied to test the associations among variables. Multiple logistic regression analysis was performed to assess the relationship between the genotype of patients (NAFLD treated wild type vs mutated patients) and the therapeutic outcome on: insulin, HOMA-IR, ALT, CRP and TBARS. The investigators identified in the following values the specific cut-offs to consider the parameter improved: insulin normalization (< 24 micro-IU/ml), normalization of the HOMA-IR (<2.5) at the end of treatment starting from baseline values greater than 2.5 and/or reduction of the HOMA-IR ≥ 2 points at the end of treatment in comparison to baseline, ALT normalization (<45 IU/L), CRP normalization (<0.6 mg/dL) or reduction of at least 1 mg/dL, TBARS reduction of at least 10 nmol/μg. The abovementioned parameters were chosen in relation to the main therapeutic effect of silybin in this context, considering NAFLD as a systemic disease. The relative risk (RR) of a useful therapeutic outcome considering the genotype of the patients was calculated considering the confounding variables (age, sex, comorbidities, medications, liver stiffness and CAP). Statistical significance was defined as p<0.05 in a two-tailed test with a 95% Confidence Interval.

Statistical analyses were performed using Statistical Program for Social Sciences (SPSS®) vs.18.0.

ELIGIBILITY:
Inclusion criteria

* age between 18 and 80 years
* diagnosis of NAFLD

Exclusion criteria

* diagnosis of chronic inflammatory disease such as inflammatory bowel disease, rheumatoid arthritis, acute or chronic kidney disease, systemic lupus erythematosus, or other major inflammatory systemic diseases
* diagnosis of insulin dependent diabetes
* diagnosis of tumors
* diagnosis of ongoing infections
* alcohol or drug abuse medical history
* diagnosis of other etiologies of chronic liver damage
* use of hepatoprotective drugs
* psychological/psychiatric problems that could invalidate the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Number of participants in each study group which shown an improvement from baseline of insulin resistance assed by HOMA-IR | Six months
  The HOMA-IR was calculated using the following formula: fasting insulin (μU/mL) × plasma glucose (mmol/L)/22.5. The investigators considered the patients responder if at least one of the following criteria was addressed: normalization of the HOMA-IR (<2.5) at the end of treatment starting from baseline values greater than 2.5; reduction of the HOMA-IR ≥ 2 points at the end of treatment in comparison to baseline.

SECONDARY OUTCOMES:
Mean change in ALT levels from baseline | Six months
  The ALT levels were assessed using a colorimetric commercially available kits and expressed as IU/L. The investigators also considered the parameter improved from the baseline in case of normalization (<45 IU/L).
Mean change in insulin levels from baseline | Six months
  The insulin levels were measured enzymatically using commercially available kits and expressed as micro-IU/ml. The investigators also considered the parameter improved from the baseline in case of normalization (<24 micro-IU/ml).
Mean change in CRP levels from baseline | Six months
  The CRP levels were measured enzymatically using commercially available kits and expressed as mg/dl. The investigators also considered the parameter improved from the baseline in case of CRP normalization (<0.6 mg/dL) or reduction of at least 1 mg/dL.
Mean change in TBARS levels from baseline | Six months
  TBARS assay was performed using 10 μl of serum. The cromogen TBARS was quantified using a spectrophotometer at a wavelength of 532nm with 1,1,3,3-tetramethoxyprophane as a standard. The amount of TBARS was expressed as nmol/μg of protein. The investigators also considered the parameter improved from the baseline in case of TBARS reduction of at least 10 nmol/μg

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Federico, Professor, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (3):
- Italy (3):
  - University of Salerno, Fisciano, Salerno
  - University of Campania "Luigi Vanvitelli", Naples
  - University of Naples "Federico II), Naples

IPD SHARING:
Plan to Share IPD: Yes
All the data that underlie results in a publication are available for the IPD sharing process upon reasonable request to the principal investigator.
  The access to the data will be granted to Researchers who provide a methodologically sound proposal. Proposals should be directed to alessandro.federico@unicampania.it or marcello.dallio@unicampania.it. To gain access, data requestors will need to sign a data access agreement. Data are available starting 6 months after publication for 10 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication for 10 years
Access Criteria: All the data that support the results of the publication will be shared upon reasonable request by correspondence to alessandro.federico@unicampania.it or marcello.dallio@unicampania.it

REFERENCES:
- [Background] Lu FB, Zheng KI, Rios RS, Targher G, Byrne CD, Zheng MH. Global epidemiology of lean non-alcoholic fatty liver disease: A systematic review and meta-analysis. J Gastroenterol Hepatol. 2020 Dec;35(12):2041-2050. doi: 10.1111/jgh.15156. Epub 2020 Jul 7. PMID 32573017
- [Background] Harris R, West J, Morling JR. Editorial: how widespread and serious is non-alcoholic fatty liver disease in the real world? Aliment Pharmacol Ther. 2020 Jun;51(11):1199-1200. doi: 10.1111/apt.15714. No abstract available. PMID 32424922
- [Background] Dallio M, Masarone M, Errico S, Gravina AG, Nicolucci C, Di Sarno R, Gionti L, Tuccillo C, Persico M, Stiuso P, Diano N, Loguercio C, Federico A. Role of bisphenol A as environmental factor in the promotion of non-alcoholic fatty liver disease: in vitro and clinical study. Aliment Pharmacol Ther. 2018 Mar;47(6):826-837. doi: 10.1111/apt.14499. Epub 2018 Jan 11. PMID 29322544
- [Background] Nicolucci C, Errico S, Federico A, Dallio M, Loguercio C, Diano N. Human exposure to Bisphenol A and liver health status: Quantification of urinary and circulating levels by LC-MS/MS. J Pharm Biomed Anal. 2017 Jun 5;140:105-112. doi: 10.1016/j.jpba.2017.02.058. Epub 2017 Mar 10. PMID 28346880
- [Background] Marchesini G, Bugianesi E, Forlani G, Cerrelli F, Lenzi M, Manini R, Natale S, Vanni E, Villanova N, Melchionda N, Rizzetto M. Nonalcoholic fatty liver, steatohepatitis, and the metabolic syndrome. Hepatology. 2003 Apr;37(4):917-23. doi: 10.1053/jhep.2003.50161. PMID 12668987
- [Background] Federico A, Dallio M, Caprio GG, Ormando VM, Loguercio C. Gut microbiota and the liver. Minerva Gastroenterol Dietol. 2017 Dec;63(4):385-398. doi: 10.23736/S1121-421X.17.02375-3. PMID 28927250
- [Background] Santoro N, Kursawe R, D'Adamo E, Dykas DJ, Zhang CK, Bale AE, Cali AM, Narayan D, Shaw MM, Pierpont B, Savoye M, Lartaud D, Eldrich S, Cushman SW, Zhao H, Shulman GI, Caprio S. A common variant in the patatin-like phospholipase 3 gene (PNPLA3) is associated with fatty liver disease in obese children and adolescents. Hepatology. 2010 Oct;52(4):1281-90. doi: 10.1002/hep.23832. PMID 20803499
- [Background] Burza MA, Pirazzi C, Maglio C, Sjoholm K, Mancina RM, Svensson PA, Jacobson P, Adiels M, Baroni MG, Boren J, Ginanni Corradini S, Montalcini T, Sjostrom L, Carlsson LM, Romeo S. PNPLA3 I148M (rs738409) genetic variant is associated with hepatocellular carcinoma in obese individuals. Dig Liver Dis. 2012 Dec;44(12):1037-41. doi: 10.1016/j.dld.2012.05.006. Epub 2012 Jun 15. PMID 22704398
- [Background] Santoro N, Savoye M, Kim G, Marotto K, Shaw MM, Pierpont B, Caprio S. Hepatic fat accumulation is modulated by the interaction between the rs738409 variant in the PNPLA3 gene and the dietary omega6/omega3 PUFA intake. PLoS One. 2012;7(5):e37827. doi: 10.1371/journal.pone.0037827. Epub 2012 May 21. PMID 22629460
- [Background] Chalasani N, Guo X, Loomba R, Goodarzi MO, Haritunians T, Kwon S, Cui J, Taylor KD, Wilson L, Cummings OW, Chen YD, Rotter JI; Nonalcoholic Steatohepatitis Clinical Research Network. Genome-wide association study identifies variants associated with histologic features of nonalcoholic Fatty liver disease. Gastroenterology. 2010 Nov;139(5):1567-76, 1576.e1-6. doi: 10.1053/j.gastro.2010.07.057. Epub 2010 Aug 11. PMID 20708005
- [Background] Kozlitina J, Smagris E, Stender S, Nordestgaard BG, Zhou HH, Tybjaerg-Hansen A, Vogt TF, Hobbs HH, Cohen JC. Exome-wide association study identifies a TM6SF2 variant that confers susceptibility to nonalcoholic fatty liver disease. Nat Genet. 2014 Apr;46(4):352-6. doi: 10.1038/ng.2901. Epub 2014 Feb 16. PMID 24531328
- [Background] Liu YL, Reeves HL, Burt AD, Tiniakos D, McPherson S, Leathart JB, Allison ME, Alexander GJ, Piguet AC, Anty R, Donaldson P, Aithal GP, Francque S, Van Gaal L, Clement K, Ratziu V, Dufour JF, Day CP, Daly AK, Anstee QM. TM6SF2 rs58542926 influences hepatic fibrosis progression in patients with non-alcoholic fatty liver disease. Nat Commun. 2014 Jun 30;5:4309. doi: 10.1038/ncomms5309. PMID 24978903
- [Background] Mancina RM, Dongiovanni P, Petta S, Pingitore P, Meroni M, Rametta R, Boren J, Montalcini T, Pujia A, Wiklund O, Hindy G, Spagnuolo R, Motta BM, Pipitone RM, Craxi A, Fargion S, Nobili V, Kakela P, Karja V, Mannisto V, Pihlajamaki J, Reilly DF, Castro-Perez J, Kozlitina J, Valenti L, Romeo S. The MBOAT7-TMC4 Variant rs641738 Increases Risk of Nonalcoholic Fatty Liver Disease in Individuals of European Descent. Gastroenterology. 2016 May;150(5):1219-1230.e6. doi: 10.1053/j.gastro.2016.01.032. Epub 2016 Feb 2. PMID 26850495
- [Background] Federico A, Dallio M, Masarone M, Gravina AG, Di Sarno R, Tuccillo C, Cossiga V, Lama S, Stiuso P, Morisco F, Persico M, Loguercio C. Evaluation of the Effect Derived from Silybin with Vitamin D and Vitamin E Administration on Clinical, Metabolic, Endothelial Dysfunction, Oxidative Stress Parameters, and Serological Worsening Markers in Nonalcoholic Fatty Liver Disease Patients. Oxid Med Cell Longev. 2019 Oct 15;2019:8742075. doi: 10.1155/2019/8742075. eCollection 2019. PMID 31737175
- [Background] Forouhi NG, Luan J, Cooper A, Boucher BJ, Wareham NJ. Baseline serum 25-hydroxy vitamin d is predictive of future glycemic status and insulin resistance: the Medical Research Council Ely Prospective Study 1990-2000. Diabetes. 2008 Oct;57(10):2619-25. doi: 10.2337/db08-0593. Epub 2008 Jun 30. PMID 18591391
- [Background] Barchetta I, De Bernardinis M, Capoccia D, Baroni MG, Fontana M, Fraioli A, Morini S, Leonetti F, Cavallo MG. Hypovitaminosis D is independently associated with metabolic syndrome in obese patients. PLoS One. 2013 Jul 31;8(7):e68689. doi: 10.1371/journal.pone.0068689. Print 2013. PMID 23935881
- [Background] Boursier J, Zarski JP, de Ledinghen V, Rousselet MC, Sturm N, Lebail B, Fouchard-Hubert I, Gallois Y, Oberti F, Bertrais S, Cales P; Multicentric Group from ANRS/HC/EP23 FIBROSTAR Studies. Determination of reliability criteria for liver stiffness evaluation by transient elastography. Hepatology. 2013 Mar;57(3):1182-91. doi: 10.1002/hep.25993. Epub 2013 Feb 4. PMID 22899556
- [Background] Sasso M, Miette V, Sandrin L, Beaugrand M. The controlled attenuation parameter (CAP): a novel tool for the non-invasive evaluation of steatosis using Fibroscan. Clin Res Hepatol Gastroenterol. 2012 Feb;36(1):13-20. doi: 10.1016/j.clinre.2011.08.001. Epub 2011 Sep 15. PMID 21920839
- [Background] Uchida D, Takaki A, Oyama A, Adachi T, Wada N, Onishi H, Okada H. Oxidative Stress Management in Chronic Liver Diseases and Hepatocellular Carcinoma. Nutrients. 2020 May 28;12(6):1576. doi: 10.3390/nu12061576. PMID 32481552
- [Background] Loguercio C, Andreone P, Brisc C, Brisc MC, Bugianesi E, Chiaramonte M, Cursaro C, Danila M, de Sio I, Floreani A, Freni MA, Grieco A, Groppo M, Lazzari R, Lobello S, Lorefice E, Margotti M, Miele L, Milani S, Okolicsanyi L, Palasciano G, Portincasa P, Saltarelli P, Smedile A, Somalvico F, Spadaro A, Sporea I, Sorrentino P, Vecchione R, Tuccillo C, Del Vecchio Blanco C, Federico A. Silybin combined with phosphatidylcholine and vitamin E in patients with nonalcoholic fatty liver disease: a randomized controlled trial. Free Radic Biol Med. 2012 May 1;52(9):1658-65. doi: 10.1016/j.freeradbiomed.2012.02.008. Epub 2012 Feb 15. PMID 22343419
- [Background] Federico A, Trappoliere M, Tuccillo C, de Sio I, Di Leva A, Del Vecchio Blanco C, Loguercio C. A new silybin-vitamin E-phospholipid complex improves insulin resistance and liver damage in patients with non-alcoholic fatty liver disease: preliminary observations. Gut. 2006 Jun;55(6):901-2. doi: 10.1136/gut.2006.091967. No abstract available. PMID 16698763
- [Background] Trappoliere M, Caligiuri A, Schmid M, Bertolani C, Failli P, Vizzutti F, Novo E, di Manzano C, Marra F, Loguercio C, Pinzani M. Silybin, a component of sylimarin, exerts anti-inflammatory and anti-fibrogenic effects on human hepatic stellate cells. J Hepatol. 2009 Jun;50(6):1102-11. doi: 10.1016/j.jhep.2009.02.023. Epub 2009 Apr 5. PMID 19398228
- [Derived] Dallio M, Masarone M, Romeo M, Tuccillo C, Morisco F, Persico M, Loguercio C, Federico A. PNPLA3, TM6SF2, and MBOAT7 Influence on Nutraceutical Therapy Response for Non-alcoholic Fatty Liver Disease: A Randomized Controlled Trial. Front Med (Lausanne). 2021 Oct 8;8:734847. doi: 10.3389/fmed.2021.734847. eCollection 2021. PMID 34692725